CLINICAL TRIAL: NCT02755142
Title: Clinical Phase I/II Study on 5-aminolevulinic Acid Hydrochloride (5-ALA) for Fluorescence-guided Resection of Malignant Gliomas
Brief Title: Clinical Study on 5-aminolevulinic Acid Hydrochloride (5-ALA) for Fluorescence-guided Resection of Malignant Gliomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: medac GmbH (Industry)
Collaborators: IKP (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: MC-ALS.8-I/GLI
Record Dates: First submitted 2016-04-22; First posted 2016-04-28 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-04

CONDITIONS: Brain Neoplasm
MeSH Terms: conditions — Brain Neoplasms | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose level 1 (Active Comparator): 0,2 mg/Kg
  Interventions: Biological: Gliolan
- Dose level 2 (Active Comparator): 2,0 mg/Kg
  Interventions: Biological: Gliolan
- Dose level 3 (Active Comparator): 20 mg/Kg
  Interventions: Biological: Gliolan

INTERVENTIONS:
Biological: Gliolan
  Other Names: 5-Aminolevulinic Acid Hydrochloride (5-ALA)

SUMMARY:
This study is planned to detect a dose-efficacy relationship between the chosen dose levels of MC506/1 and the extent and quality of fluorescence in the tumour core in patients with newly diagnosed malignant glioma.

ELIGIBILITY:
Inclusion Criteria:

* Radiological suspicion of a malignant glioma with distinct ring- or garland shaped, contrast agent-enhancing tumour structures and a core area of reduced intensity in the MRI (tumour necrosis)
* Indication for surgical tumour resection
* First operation of the tumour, no other tumour-specific pre-treatment
* Karnofsky Performance Scale 70%
* Patient's written informed consent
* Age 18-75 years

Exclusion Criteria:

* Porphyria, hypersensitivity to porphyrins
* Renal insufficiency:

  * Creatinine > 2.0 mg/dl
* Hepatic insufficiency:

  * Bilirubin > 3 mg/dl
  * Quick test < 60 %
  * GT > 100 U/I
* Other known malignancy (except basaliomas)

Women:

* Existing/planned pregnancy (to be checked by a pregnancy test if of child-bearing age)/lactation or inadequate contraception (hormone cycle regulation pill or condom)

Men:

* Inadequate contraception (condom)
* Dementia or mental condition making it impossible to understand the therapy and therefore prohibiting written consent
* Simultaneous participation or participation in another clinical trial in the preceding 30 days

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2000-02; Primary Completion 2001-06 (Actual); Study Completion 2001-06 (Actual)

PRIMARY OUTCOMES:
Detection of a dose-efficacy relationship between the dose levels and the extent and quality of fluorescence in the tumour core (of newly diagnosed malignant glioma). | Within 3 hours
  After completion of resection, global fluorescence extent in the tumour core will be assessed by the first and second surgeon. It will be estimated whether approx. 0/3, 1/3, 2/3 or 3/3 of the tumour core is identified using standard white operation light were fluorescent (irrespective of fluorescence quality). The global quality of Gliolan induced tissue fluorescence within the tumour core will be recorded as being strong, weak or missing. As an objective control of the subjective assessment of the fluorescent quality, selected areas will be measured spectrometrically.

IPD SHARING:
Plan to Share IPD: No